CLINICAL TRIAL: NCT04827303
Title: Effectiveness of 3 Different Methods in Acute Myofascial Pain Syndrome: A Randomized Controlled Study
Brief Title: Effectiveness of Different Methods in Acute Myofascial Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Saime Ay, Professor Doctor, Ufuk University
Other Study IDs: 29032017-8
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Myofacial Pain Syndromes
MeSH Terms: conditions — Facial Neuralgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Kinesio taping — A 10-15 cm sized I band was applied to the trapezius muscles of the first group patients with the patient's neck in lateral flexion. Then, while the patient's neck is flexed, a Y-shaped 15-20 cm tape will be affixed between C1-7 with the arms of the Y up, and I tape of 5-10 cm is attached on the arms. In group 2 patients, 1 cc lidocaine diluted with 4 cc saline (SF) was applied to the trigger points palpated manually in the trapezius muscles. After the trigger point was squeezed between the thumb and index finger, a few cc of local anesthetic mixture was applied into the trigger point with the injector and exited. In the 3rd group patients, a few cc local anesthetic mixture will be applied intradermally over the trigger point without entering into the trigger points palpated manually in the trapezius muscles. Patients were checked 72 hours and 1 week after the first applications.
  Other Names: trigger point injection; neural therapy injection

SUMMARY:
This study is a randomized controlled study. A total of 75 patients between the ages of 20-50 who have a diagnosis of acute myofacial pain syndrome in the trapezius muscle and have pain for a maximum of 5 days were included in the study. Patients were randomly divided into 3 groups. Group 1 patients received kinesio tape method (25 patients), group 2 patients received trigger point injection method (25 patients), and group 3 patients received neural therapy injection method (25 patients). A 10-15 cm sized I band was applied to the trapezius muscles of the first group patients with the patient's neck in lateral flexion. Then, while the patient's neck is flexed, a Y-shaped 15-20 cm tape will be affixed between C1-7 with the arms of the Y up, and I tape of 5-10 cm is attached on the arms. In group 2 patients, 1 cc lidocaine diluted with 4 cc saline (SF) was applied to the trigger points palpated manually in the trapezius muscles. After the trigger point was squeezed between the thumb and index finger, a few cc of local anesthetic mixture was applied into the trigger point with the injector and exited. In the 3rd group patients, a few cc local anesthetic mixture will be applied intradermally over the trigger point without entering into the trigger points palpated manually in the trapezius muscles. Patients were checked 72 hours and 1 week after the first applications.

The pain at rest and during movement of the patients in all 3 groups were evaluated with a visual analog scale (VAS 10 cm). The number of trigger points was determined by the physician by hand palpation. Pressure pain threshold was evaluated with the algometer device. Disability assessment of the patients was made using the neck pain disability index. evaluations were made at the beginning of treatment, 72 hours after and 1 week after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute myofascial pain syndrome
* Patients between the ages of 20-50
* Patients with pain for up to 5 days

Exclusion Criteria:

* Patients diagnosed with fibromyalgia
* Patients with systemic disease
* Patients with prominent cervical disc herniation
* Patients with cervical arthrosis
* Patients with cervical radiculopathy and myelopathy
* Patients with myofascial trigger point injection in the past 6 months
* Patients who received physical therapy in the past 6 months
* Patients undergoing shoulder and neck surgery
* Patients with drug allergies

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 75 patients between the ages of 20-50 who have a diagnosis of acute myofacial pain syndrome in the trapezius muscle and have pain for a maximum of 5 days.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 1 week
  The pain at rest and during movement of the patients in all 3 groups were evaluated with a visual analog scale (VAS 10 cm).
The number of trigger points | 1 week
  The number of trigger points was determined by the physician by hand palpation.
Pressure pain threshold | 1 week
  Pressure pain threshold was evaluated with the algometer device.
Neck pain disability index | 1 week
  Disability assessment of the patients was made using the neck pain disability index.

CONTACTS AND LOCATIONS:
Overall Officials: saime ay, Principal Investigator — Ufuk University
Locations (1):
- Ufuk University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided